CLINICAL TRIAL: NCT02442323
Title: A Pilot Study of a Home-Based Walking Intervention for Pancreatic Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Principal Investigator, Carolyn Fang, PhD, Principal Investigator, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB13023
Record Dates: First submitted 2015-03-18; First posted 2015-05-13 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking Intervention (Experimental): Intervention patients will receive a 12-week home-based walking program, which includes a personalized instruction booklet and pedometer. The walking program consists of 3 phases and will be individualized for each patient based on their physical condition and baseline assessment. Patients are instructed to walk 3 to 5 times each week at home or other safe environment. Patients will be instructed on a gradual increase in walking time over the course of the intervention.
  Interventions: Behavioral: Walking Intervention
- Usual Care (No Intervention): Usual care patients will receive standard of care. They will not receive any instruction on walking or other physical activity other than what is normally provided by their physician or clinical staff.

INTERVENTIONS:
Behavioral: Walking Intervention — 12-week walking program
  Arms: Walking Intervention

SUMMARY:
Despite evidence regarding the benefits of physical activity in various cancer patient populations, the effects of a home-based walking program for pancreatic cancer patients have been under-explored. The aims of the proposed pilot project are to: (1) Assess the feasibility of implementing a 12-week, home-based walking program among pancreatic cancer patients; and (2) Examine the effects of a 12-week, home-based walking program on quality of life (QOL) and symptoms among pancreatic cancer patients.

DETAILED DESCRIPTION:
Among cancer patients, physical activity interventions can lead to improvements in QOL and reductions in fatigue and pain. While pancreatic cancer patients may have physical restrictions that limit their participation in moderate to high-intensity exercise activities, empirical evidence suggests that even low-intensity, home-based walking programs can confer benefits for cancer patients. In this pilot study, 50 patients will be randomly assigned to receive either the walking intervention program or usual care (UC). Assessments of quality of life, distress, and symptom burden will be completed at baseline (pre-intervention) and at follow-up (i.e. within 2 weeks post-intervention or approximately 12-14 weeks post-baseline). Data from the proposed pilot study will inform the development of a larger randomized trial designed to improve QOL and reduce morbidity in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Have histologically confirmed adenocarcinoma of the pancreas (including adenocarcinoma subtypes such as signet ring carcinoma, adenosquamous carcinoma, undifferentiated/poorly differentiated carcinoma, and mucinous carcinoma)
* Have an estimated life expectancy of greater than 3 months
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Are undergoing treatment for pancreatic cancer at Fox Chase Cancer Center
* Have borderline resectable or unresectable locally advanced disease or metastatic disease

Exclusion Criteria:

* Patients with islet cell/neuroendocrine or papillary cystic neoplasm
* Patients scheduled to undergo surgical resection for curative intent during study participation
* Patients receiving 3rd-line palliative chemotherapy
* Inability to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported outcome of quality of life | 14 weeks post-baseline
  Quality of life will be measured using the FACT-Hep, a validated tool that assesses 4 components of quality of life (physical well-being, emotional well-being, social well-being, and functional well-being), as well as common symptoms associated with hepatobiliary cancers, including pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y Fang, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States